CLINICAL TRIAL: NCT00314704
Title: Comparison of Dopamine and Norepinephrine as the First Vasopressor Agent in the Management of Shock
Brief Title: Dopamine and Norepinephrine in Shock Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sepsis Occurrence in Acutely Ill Patients (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOAP vasopressors
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2006-04

CONDITIONS: Shock
Keywords: shock; hypotension; circulatory failure; septic shock; cardiogenic shock
MeSH Terms: conditions — Shock; Hypotension; Shock, Septic; Shock, Cardiogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: dopamine versus norepinephrine

SUMMARY:
The purpose of this study is to compare the efficacy of dopamine and norepinephrine, two commonly used vasopressor agents, in the treatment of shock.

DETAILED DESCRIPTION:
Introduction:

Vasopressor agents are commonly used to correct hypotension in patients with acute circulatory failure. Their variable alpha, beta, or dopaminergic receptor stimulation, may result in different hemodynamic and metabolic effects. Several experimental and human studies have indicated that dopamine and norepinephrine may have different effects on the kidney, the splanchnic region or the pituitary axis, but the implications of these findings have not been assessed. Hence, both agents are widely used, and several consensus or expert recommendations still recommend the use of both agents 1,2. An observational study has reported that dopamine and epinephrine may be associated with a higher mortality rate than norepinephrine 3. In addition, The results of the SOAP study indicated that dopamine may be associated with higher mortality rates than norepinephrine, but various uncontrolled factors may have influenced these results. Therefore, we will address this issue in a prospective, randomized, double blind study. We hypothesize that both agents have similar effects on survival.

Design of the study:

Prospective, randomized, double blind, multicenter.

Patients:

A total of 1600 consecutive patients with hypotension requiring the administration of vasopressors.

Power calculation: Calculation is based on the results of the SOAP study (mortality 43% with dopamine and 36% with norepinephrine), using a two-sided analysis, with a significant p value at 0.05 and a power of 80%, 765 patients are needed in each group. About 40 centers will be recruited.

Inclusion criteria:

Mean arterial pressure less than 70 mmHg or systolic pressure less than 100 mmHg persisting despite adequate fluid loading (in example with at least 1000 mL crystalloid or 500 ml colloid) unless central venous pressure (CVP) or pulmonary artery occluded pressure (PAOP) are elevated (e.g. CVP> 12 mmHg or PAOP > 14 mmHg).

Exclusions:

* Serious arrhythmia such as rapid atrial fibrillation (> 160/min) or ventricular tachycardia.
* Brain death.
* Open label administration of dopamine, norepinephrine, epinephrine or phenylephrine for more than 4hours.

Consent:

Patients will be randomized immediately, with the use of sealed envelopes placed near the supplies of dopamine and norepinephrine. If the patient is already being treated with one agent, randomization can still take place provided that it is within a 4 hour period.

Consent will be obtained from the patient before entering the study, if possible, or from the next of kin as soon as possible after starting vasopressor therapy. Indeed, in such cases, vasopressor therapy should anyway be started, either with dopamine or with norepinephrine, and these 2 therapies are currently equally valid 1st choices. As soon as possible, the next of kin will be informed and deferred consent obtained. If the patient recovers, and is able to consent, consent will then be obtained.

According to local Ethical Committee, oral or signed consents will be obtained.

Protocol:

Blood pressure goal: defined by the physician in charge, according to each unit's recommendations

Administration of vasoactive drugs:

Double blind administration of a solution of norepinephrine or dopamine contained either in vials or syringes according to the ICU's protocol (see appendices I and II for vial and syringe preparations). Each solution will be labeled with its randomly allocated number and will be prepared by the nurses in charge. The rate of administration of the blind solution will be determined according to a scale and using the estimated body weight. The recommended steps for increasing or decreasing the doses of the blinded solution are calculated to be equivalent to 2 µg/kg.min for dopamine and 0.02 mcg/kg.min for norepinephrine, the investigator being free to use multiples of this increment in case of emergency. The maximal dose with the 2 agents will be 20 µg/kg.min for dopamine and 0.19 mcg/kg.min for norepinephrine (these doses have been shown to have similar effects on mean arterial blood pressure 4).

If the patient is already treated with open label vasopressors at baseline, the blinded solution will be rapidly incremented, and, if possible, the open label vasopressor agent will be decreased. If this open label vasopressor consisted in dopamine and if this agent cannot be fully weaned after the introduction of the blinded solution, the open label dopamine will be replaced by an open label norepinephrine infusion.

When the maximal dose of the blinded solution is achieved, an open label perfusion of norepinephrine can be added to achieve the desired blood pressure. Epinephrine or vasopressin may be used only as rescue therapy. Weaning of vasopressor agents will begin by weaning of the open label norepinephrine, followed by weaning of the blinded solution. In case of recurrence of hypotension, the blinded solution will be resumed first (maximal dose with the 2 agents will be 20 µg/kg.min for dopamine and 0.19 mcg/kg.min for norepinephrine) and if needed an open label solution of norepinephrine may be added. Weaning of the vasopressors will be performed as previously described.

Dobutamine, dopexamine, and inhibitors of phosphodiesterase III can be used, if needed, to optimize cardiac output according to local practices.

General therapeutic guidelines:

All therapies will be performed according to local guidelines. The choice of sedative agents, antibiotics, fluids, transfusion threshold, ventilatory modes,…. , will be left to the attending physicians. Likewise, the administration of agents like corticosteroids or drotrecogin-alpha activated (Xigris) is permitted.

Randomization:

Randomization by blocks for each participating ICU, using a computer generated list to allocate treatments A or B, put in sealed envelopes near the drug supplies. In each ICU, sealed envelopes including treatment allocation and a five digit number will be available. The envelope will be opened by the person responsible for preparation of the dopamine and norepinephrine solutions. The random number and treatment allocation will be written on a hidden book, available only for the person responsible for preparation of the dopamine and norepinephrine solutions. The doctors and other nurses will be kept blinded to treatment allocation. On patients' charts only the rate of administration and the dilution (simple or double) of the solution will be written.

Preparation of the solutions:

The solutions of dopamine or norepinephrine will be prepared by the nurse in charge of the patient. The five digit number (allocated by randomization) will be written on the bag. See appendices I and II for details regarding the preparation of the solutions. Different concentrations of these solutions are provided, the choice of the concentration of the solution will be left to the physician in charge.

Definition of the end of the shock period:

Shock will be considered as having resolved when the investigational drug can be stopped for more than 12 hours.

End-points:

Primary end-point: 28 day survival

Secondary end-points:

ICU survival Hospital survival Severity of organ dysfunction in the ICU (SOFA score 5) Duration of ICU stay, time spent on vasopressors (vasopressor free days), on mechanical ventilation (ventilator free days) and on renal replacement (renal replacement free days) Efficacy of dopamine to correct hypotension Hemodynamic effects / concomitant use of dobutamine or other inotropic agents Tolerance: arrhythmia (incidence of ventricular tachycardia, ventricular fibrillation and atrial fibrillation), myocardial necrosis, skin necrosis, limb or distal extremity ischemia.

Occurrence of secondary infections Impact of target blood pressure on outcome

Measured variables:

Data to be collected every 6 hours for 48 hours and then every 8 hours up to day 5

Hemodynamic variables:

Temperature, systolic and diastolic arterial pressures, heart rate, central venous pressure.

In patients equipped with a pulmonary artery catheter: pulmonary systolic and diastolic pressures, pulmonary artery occluded pressure, cardiac output.

In patients equipped with devices allowing cardiac output measurement: cardiac output, extravascular lung water and global end diastolic volumes (if available)

Biologic variables:

Arterial and mixed-venous (or central venous if pulmonary artery catheter not available) blood gases.

Doses of vasoactive agents: trial drug, open label vasoactive drugs (norepinephrine, epinephrine, vasopressin, dobutamine)

Data to be collected daily for the first 7 days and then on days 14, 21 and 28:

Hemoglobin, platelets, white blood cell count, APTT, glucose levels, urea, creatinine, sodium, potassium, GOT, GPT, CPK, LDH, PAL, bilirubin, amylase, lipase, CRP, lactate, PCT (if available) Respiratory conditions (type of ventilation and condition) Fluid balance (In/Out) Microbiological data and antibiotic therapy

Calculation of APACHE II 6 and SAPS II scores on admission and on inclusion in the study and calculation of SOFA score daily for the first 7 days and then on days 14, 21 and 28.

Statistics:

A/ Interim analysis: Sequential analysis every 100 included patients, allowing premature stop of the study in case of significant difference in 28-day survival between the two treatments, or futility

B/ Final analysis:

Intention to treat analysis Kaplan-Meier curves (with log rank test) will be used to assess ICU and 28-day survival as well as the durations of vasopressor therapy (both for labeled and open label drugs) and ICU stay.

Analysis of variance followed by t-test with Bonferroni correction for all continuous variables and chi square for categorial variables.

Significance at p< 0.05.

C/ Additional and subgroup analysis:

* Analysis of subgroup is scheduled for septic shock, cardiogenic shock, and all other types of shock.
* Per protocol analysis, to take into account patients excluded for arrhythmias.
* Subgroup analysis according to the dose of vasoactive agents (trial drug only and trial plus open label drugs)

References:

1. Task Force of the American College of Critical Care Medicine, Society of Critical Care Medicine. Practice parameters for hemodynamic support of sepsis in adult patients in sepsis. Crit Care Med 1999; 27:639-660.
2. Vincent J-L. Hemodynamic support in septic shock. Intensive Care Med 2001; 27:S80-S92
3. Martin C, Viviand X, Leone M, Thirion X. Effect of norepinephrine on the outcome of septic shock. Crit Care Med 2000; 28:2758-2765.
4. Marik PE, Mohedin M. The contrasting effects of dopamine and norepinephrine on systemic and splanchnic oxygen utilization in hyperdynamic sepsis. JAMA 1994; 272:1354-1357.
5. Vincent JL, Moreno J, Takala J, Willatts S, De Mendonça A, Bruining H, et al. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. Intensive Care Med 2000; 22:707-710.
6. Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med 1985; 13:818-829.

ELIGIBILITY:
Inclusion Criteria:

* Mean arterial pressure less than 70 mmHg or systolic pressure less than 100 mmHg persisting despite adequate fluid loading (in example with at least 1000 mL crystalloid or 500 ml colloid) unless central venous pressure (CVP) or pulmonary artery occluded pressure (PAOP) are elevated (e.g. CVP> 12 mmHg or PAOP > 14 mmHg).

Exclusion Criteria:

* Serious arrhythmia such as rapid atrial fibrillation (> 160/min) or ventricular tachycardia.
* Brain death.
* Open label administration of dopamine, norepinephrine, epinephrine or phenylephrine for more than 4hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1679 (Actual)
Dates: Start 2003-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
28 day survival

SECONDARY OUTCOMES:
ICU survival
Hospital survival
Severity of organ dysfunction in the ICU (SOFA score)
Duration of ICU stay
Time spent on vasopressors (vasopressor free days)
Time spent on mechanical ventilation (ventilator free days)
Time spent on renal replacement (renal replacement free days)
Efficacy of dopamine to correct hypotension
Hemodynamic effects
Concomitant use of dobutamine or other inotropic agents
Tolerance: arrhythmia (incidence of ventricular tachycardia, ventricular fibrillation and atrial fibrillation), myocardial necrosis, skin necrosis, limb or distal extremity ischemia.
Occurrence of secondary infections
Impact of target blood pressure on outcome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel De Backer, MD, PhD, Principal Investigator — SOAP investigators
Locations (8):
- University Hospital of Vienna, Vienna, Austria
- Belgium (6):
  - CHU Saint Pierre, Brussels
  - CHU Brugmann, Brussels
  - HIS Ixelles, Brussels
  - Erasme University Hospital, Brussels
  - St Elisabeth, Brussels
  - CHU Charleroi, Charleroi
- Hospital Universitario Rio Hortega, Valladolid, Spain

REFERENCES:
- [Derived] De Backer D, Biston P, Devriendt J, Madl C, Chochrad D, Aldecoa C, Brasseur A, Defrance P, Gottignies P, Vincent JL; SOAP II Investigators. Comparison of dopamine and norepinephrine in the treatment of shock. N Engl J Med. 2010 Mar 4;362(9):779-89. doi: 10.1056/NEJMoa0907118. PMID 20200382
- See also: Click here for more information about this study: Dopamine and norepinephrine as the first vasoactive agent — http://www.intensive.org